CLINICAL TRIAL: NCT06035120
Title: An Evaluation of the AeriSeal System for CONVERTing Collateral Ventilation Status in Patients With Severe Emphysema: The CONVERT II Trial
Brief Title: An Evaluation of the AeriSeal System for CONVERTing Collateral Ventilation Status in Patients With Severe Emphysema
Acronym: CONVERT_II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 630-2000-01
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Emphysema, Pulmonary; Emphysema or COPD
Keywords: Collateral Ventilation; Bronchoscopic Lung Volume Reduction; Hyperinflation
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-arm clinical trial in which eligible subjects with an identified fissure gap in the target lobe will be treated with the AeriSeal System to determine the rate of conversion from having collateral ventilation (CV+) to having little to no collateral ventilation (CV-). Subjects who convert to CV- status with AeriSeal will then undergo BLVR using Zephyr Valve per standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AeriSeal (Experimental): All enrolled subjects meeting final eligibility will undergo the AeriSeal procedure to block collateral ventilation by closing the lobar fissure gaps or collateral air channels.
  Interventions: Device: AeriSeal System

INTERVENTIONS:
Device: AeriSeal System — The AeriSeal System comprises AeriSeal Foam and the AeriSeal Balloon Catheter Preparation Kit that is used for bronchoscopic delivery of AeriSeal Foam to the targeted regions of the lung.

SUMMARY:
This is a prospective, open-label, multi-center, single-arm study planned to enroll 200 subjects with heterogeneous emphysema and collateral ventilation (CV) in the target lobe. Subjects will undergo instillation of AeriSeal Foam in the target lobe and subsequent assessment of CV status using Chartis Pulmonary Assessment System. Subjects with CV- status will then undergo placement of Zephyr Valve in the target lobe for bronchoscopic lung volume reduction (BLVR) and be followed for 24 months.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm, pivotal trial with a 24-month follow-up to evaluate the safety and effectiveness of the AeriSeal System to block CV. The study plans to enroll up to 200 subjects at up to 35 clinical centers in US and OUS. Study subjects will be patients with severe, heterogeneous emphysema and collateral ventilation in the lobe targeted who are candidates for BLVR. Subjects meeting initial eligibility will undergo a bronchoscopy procedure under general anesthesia during which the presence of CV will be confirmed using Chartis. All enrolled subjects meeting final eligibility will undergo the AeriSeal procedure. Conversion of collateral ventilation status from CV+ to CV- in the target lobe will be evaluated by Chartis at Day 45 post-AeriSeal treatment (primary effectiveness endpoint). All subjects not converted from CV+ to CV- status will undergo a repeat of the AeriSeal procedure, provided that the total volume from both the initial and the repeat treatments does not exceed 40 mL in up to 3 segments. All subjects converted from CV+ to CV- status after either the index or repeat AeriSeal procedure will undergo BLVR with Zephyr Valve per standard of care in accordance with the approved instructions for use and will be followed through Month 24 (end of study). All CV+ subjects who remain CV+ after the repeat procedure or do not undergo the repeat AeriSeal procedure will be followed through Month 24 (end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent and to participate in the study.
2. Subject is aged ≥ 40 and ≤ 80 years at the time of the ICF signature date.
3. Subject has completed a documented pulmonary rehabilitation (in clinic or home-based) program within 12 months prior to Baseline.
4. Subject has stopped smoking for at least 8 weeks prior to the ICF signature date as confirmed by carboxyhemoglobin or cotinine levels.
5. Subject has a recent HRCT meeting the scan parameter requirements and performed within 3 months of the ICF signature date with the following findings at -910 Hounsfield Units:

   1. At least one (1) lobe with segmental emphysema destruction score ≥ 50%.
   2. Subject has heterogenous emphysema, defined as difference in emphysema destruction score of ≥ 15 between the density scores of the target lobe and the ipsilateral non-target lobe(s) per QCT report with % voxel density of < -910 HU. For non-target lobes that include the RML, calculate the combination of non-target lobes as a single density score using volume-weighted percent.
   3. LUL, LLL, RUL, RLL, or RUL+RML are targets for valve intervention.
   4. Subject has a gap in the interlobar fissure that corresponds to one or more segments and the fissure(s) contacting the target lobe is ≥ 80% complete per QCT report.
   5. Subject has 98% of the fissure gap confined to a maximum of 3 segments within the target lobe per Fissure Targeting Report (FTR).
6. Subject has 6MWD ≥ 150 m and ≤ 450 m.
7. Subject has clinically significant dyspnea with an mMRC score of ≥ 2.
8. Subject has post-bronchodilation FEV1 ≥ 15% predicted and ≤ 45% predicted.
9. Subject has an FEV1/FVC ratio of < 0.7.
10. Subject has post-bronchodilation TLC, measured by body plethysmography, ≥ 100% predicted.
11. Subject has post-bronchodilation RV ≥ 175% predicted, measured by body plethysmography.
12. Subject has post-bronchodilation DLCO ≥ 20% predicted.
13. Subject has received preventative vaccinations against potential respiratory infections, including COVID-19, consistent with local recommendation or policy.
14. Subject is on optimal medical management for more than one month prior to the ICF signature date.
15. Subject has collateral ventilation (CV+) as confirmed per the Chartis assessment prior to the AeriSeal Index Procedure.

Exclusion Criteria:

1. Subject has prior lung volume reduction surgery, lobectomy or pneumonectomy, lung transplantation, airway stent placement, pleurodesis, or BLVR of any type, except BLVR using Zephyr Valve with < 50% TLVR at 6 months, followed by valve removal > 6 months prior to ICF signature date.
2. Subject has visible radiological abnormality on HRCT scan such as pulmonary nodule greater than 0.8 cm in diameter (does not apply, if present for 2 years or more without increase in size or if deemed benign by biopsy) or active pulmonary infection (e.g., unexplained parenchymal infiltrate, significant interstitial lung disease or significant pleural disease).
3. Post-COVID-19 pathology on CT, including ground glass opacities with or without consolidation, adjacent pleura thickening, interlobular septal thickening, or air bronchograms.
4. Large bullae encompassing greater than 1/3 of the total lung.
5. Subject had 3 or more COPD exacerbations requiring hospitalization within 12 months preceding the ICF signature date or a COPD exacerbation requiring hospitalization within 8 weeks of the ICF signature date. Subjects may be re-considered for future enrollment.
6. Subject has asthma as their primary diagnosis.
7. Subject has chronic bronchitis (defined as greater than 4 tablespoons of sputum production per day) as their primary diagnosis.
8. Subject has clinically significant bronchiectasis.
9. Subjects with evidence of active respiratory infection should be considered for enrollment only after satisfactory resolution.
10. Subject requires invasive ventilatory support. Note: The use of Continuous Positive Airway Pressure (CPAP) or BiPAP devices for sleep apnea is permitted.
11. Subject has severe gas exchange abnormalities as defined by any one of the following tests, conducted at rest, on room air, as tolerated.

    * PaCO2 ≥ 50 mm Hg (6.7 kPa)
    * PaO2 < 45 mm Hg (6.0 kPa)
12. Subject has pulmonary hypertension, defined as mean pulmonary systolic pressure > 45 mm Hg.
13. Subject has known documented alpha-1 antitrypsin deficiency.
14. Subject has clinically significant hematological disorder.
15. Subject has recent significant unplanned or unexplained weight loss or other relevant comorbidities considered by the investigator to be potentially confounding or limiting to the subject's participation in the study.
16. Subject has non-atrial arrhythmias or conduction abnormalities on EKG.
17. Subject has high cardiac risk after undergoing cardiac risk assessment in accordance with published guidelines (Fleisher 2007) or has ischemic heart disease, congestive heart failure, cerebrovascular disease (stroke or TIA within 6 months of the ICF signature date), serum creatinine > 2.0 mg/dL (177 μmol/L), or left ventricular ejection fraction (LVEF) < 45% on echocardiogram.
18. Subject has uncontrolled exercise induced syncope.
19. Subject has evidence of severe disease which in the judgment of the investigator may compromise the anticipated treatment effect or the subject's survival for the duration of at least 12 months.
20. Subject has any other condition that the investigator believes would interfere with the intent of the study or would make participation not in the best interest of the subject including but not limited to alcoholism, high risk for drug abuse, or noncompliance in returning for follow-up visits.
21. Subject cannot tolerate corticosteroids or relevant antibiotics.
22. Subject use of systemic corticosteroids > 20 mg/day prednisolone or equivalent within four (4) weeks of the ICF signature date. Subjects may be re-considered for future enrollment.
23. Subject use of immunosuppressive agents within four (4) weeks of the ICF signature date. Subjects may be re-considered for future enrollment.
24. Subject is unable to temporarily discontinue heparins and oral anticoagulants (e.g., warfarin, dicumarol) according to local pre-procedural protocols. Note: Antiplatelet drugs including aspirin, thienopyridines and ticagrelor are permitted.
25. Subject has allergy or sensitivity to medications required to safely perform bronchoscopy under conscious sedation or general anesthesia.
26. Subject has known allergy to the following device components: Polyether block amide (PEBAX), Polyvinyl Alcohol or Glutaraldehyde, Nitinol (nickel-titanium) or its constituent metals (nickel or titanium) or Silicone.
27. Subject is a female who is pregnant (positive βHCG Pregnancy test), breast-feeding, or planning to be pregnant in the next 12 months.
28. Subject has Body Mass Index < 18 kg/m2 or > 35 kg/m2.
29. Subject participated in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to the ICF signature date. Note: Subjects being followed as part of a long-term surveillance of a non-pulmonary study that has reached its primary endpoint are eligible for participation in this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Converters, responder rate | 45 days post-AeriSeal treatment (index or repeat)
  The percentage of study subjects that successfully convert from a positive collateral ventilation status (CV+) in the treated lobe to having little to no collateral ventilation (CV-) by Chartis.

SECONDARY OUTCOMES:
Post-bronchodilator forced expiratory volume in 1 second (FEV1), responder rate | Month 6 post-Zephyr Valve
  The percentage of converters achieving a ≥ 12% increase in FEV1
Residual volume (RV), responder rate | Month 6 post-Zephyr Valve
  The percentage of converters achieving a ≥ 310 mL decrease in RV
Treated lobe volume reduction (TLVR) by high-resolution computed tomography (HRCT), responder rate | Month 6 post-Zephyr Valve
  The percentage of converters achieving a ≥ 350 mL decrease in TLVR
St. George's Respiratory Questionnaire (SGRQ), responder rate | Month 6 post-Zephyr Valve
  The percentage of converters achieving a ≥ 4-point decrease in SGRQ total score

OTHER OUTCOMES:
Post-bronchodilator forced expiratory volume in 1 second (FEV1) change | Month 3, Month 6, Month 12, Month 24
  Absolute, percent and percent predicted change
Post-bronchodilator forced expiratory volume in 1 second (FEV1), responder rate | Month 3, Month 12, Month 24
  Percentage of subjects achieving a ≥12% increase
Residual volume (RV), responder rate | Month 3, Month 12, Month 24
  The percentage of subjects achieving a ≥ 310 mL decrease in RV
Residual volume (RV), change | Day 45, Month 6, Month 12
  Absolute and percent predicted change in RV
Treated lobe volume reduction (TLVR) by high-resolution computed tomography (HRCT), change | Day 45, Month 6, Month 12
  Absolute change in TLVR
Treated lobe volume reduction (TLVR) by high-resolution computed tomography (HRCT), responder rate | Day 45, Month 12
  The percentage of subjects achieving a ≥ 350 mL decrease in TLVR
Residual volume to total lung capacity (RV/TLC) ratio | Month 3, Month 6, Month 12, Month 24
  Absolute change in RV/TLC ratio
Forced vital capacity (FVC), change | Month 3, Month 6, Month 12, Month 24
  Absolute and percent change in FVC
Diffusion capacity of carbon monoxide (DLCO), change | Month 6, Month 12
  Absolute and percent predicted change in DLCO
Chronic Obstructive Pulmonary Disease assessment test (CAT), change | Month 3, Month 6, Month 12
  Absolute change. Minimum score: 0, maximum score: 40. Lower scores indicate a better outcome.
Chronic Obstructive Pulmonary Disease assessment test (CAT), responder rate | Month 3, Month 6, Month 12
  The percentage of subjects achieving a ≥ 2-point decrease
St. George's Respiratory Questionnaire (SGRQ), total score change | Month 3, Month 6, Month 12
  Absolute change in SGRQ total score. Minimum score: 0, maximum score: 100. Lower scores indicate a better outcome.
St. George's Respiratory Questionnaire (SGRQ), responder rate | Month 3, Month 12
  The percentage of converters achieving a ≥ 4-point decrease in SGRQ total score
Six Minute Walking Test (6MWT), responder rate | Month 6, Month 12
  Percentage of subjects achieving a ≥ 26 meter increase
Modified Medical Research Council (mMRC) Dyspnea Scale, total score change | Month 3, Month 6, Month 12
  Absolute change in total mMRC Dyspnea Scale score. Minimum score: 0, maximum score: 4. Lower scores indicate a better outcome.
Modified Medical Research Council (mMRC) Dyspnea Scale, responder rate | Month 3, Month 6, Month 12
  The percentage of subjects achieving a ≥ 1-point decrease

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Shargill, PhD, Study Director — Pulmonx Corporation
Locations (36):
- United States (18):
  - Banner University Medical Center, Phoenix, Arizona
  - Saint Francis Hospital and Medical Center (Trinity Health of New England), Hartford, Connecticut
  - Orlando Health, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham Lung Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cleveland VA Northeast, Cleveland, Ohio
  - Penn Medicine, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Fort Sanders Regional Medical Center (StatCare), Knoxville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Medical College of Wisconsin (MCW), Milwaukee, Wisconsin
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Wesley Hospital, Brisbane
  - Macquarie University, Macquarie Park
- Klinik Floridsdorf, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - CHU Limoges, Limoges
  - Hopital Bichat-APHP, Paris
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
- Germany (5):
  - Ruhrlandklink, Uni Essen, Essen
  - Universitätsklinikum Halle, Halle
  - Asklepios Klinik Barmbek, Hamburg
  - Thoraxklinik am Universitats klinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
- ASST Spedali Civili, University Hospital, Brescia, Italy
- University Medical Center Groningen, Groningen, Netherlands
- Hospital Universitario y Politecnico La Fe, Valencia, Spain
- Royal Brompton Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be aggregated and analyzed. No IPD be made available for sharing to other researchers.